CLINICAL TRIAL: NCT04763486
Title: Prophylactic Antibiotic Treatment for Perineal Tear After Delivery: a Randomized Controlled Trial
Brief Title: Prophylactic Antibiotic After Perineal Tear
Acronym: PATPET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Yair Daykan, Principal Investigator, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0189-19-MMC
Record Dates: First submitted 2019-07-29; First posted 2021-02-21 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Puerperal Infection
MeSH Terms: conditions — Puerperal Infection | interventions — Cefazolin

STUDY DESIGN:
Intervention Model Description: parturition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic antibiotic treatment (Experimental): Will be given Cefamezin antibiotic within 6 hours of delivery
  Interventions: Drug: Cefazolin (Cefamezin)
- No intervention (No Intervention): Will not get antibiotic prophylactics

INTERVENTIONS:
Drug: Cefazolin (Cefamezin) — Cefamezin 2 gr within 6 hour of delivery
  Arms: Prophylactic antibiotic treatment

SUMMARY:
Current World Health Organization guidelines recommend routine antibiotic prophylaxis for women with perineal tear 3rd and 4th degree but not for 2nd degree because of insufficient evidence of effectiveness. The investigators aimed to investigate whether antibiotic prophylaxis prevented maternal infection after the first and second perineal tear after vaginal birth.

DETAILED DESCRIPTION:
The PATPET trial is a randomized, controlled trial done at tertiary hospital obstetric units in Israel. Women who had first and second-degree tear (or after episiotomy) after delivery at 37 weeks or greater gestation, with no indication for ongoing prescription of antibiotics in the post-partum period and no contraindications to prophylactic Cefamezin (cefazolin), were randomly assigned (1:1) to receive a single intravenous dose of prophylactic antibiotic or not.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45
* perineal tear 2nd and 1st degree( episiotomy)

Exclusion Criteria:

* 3rd and 4 th degree perineal tear
* antibiotic indication during delivery
* cesarian section delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Delivery
Enrollment: 2500 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a fever after delivery | 6 weeks of delivery
  Maternal fever above 38 C (Celsius)

SECONDARY OUTCOMES:
Way of delivery | 6 weeks of delivery
  Type of delivery- vacuum-assisted delivery vs. vaginally

CONTACTS AND LOCATIONS:
Overall Officials: Gil Shechter, Dr, Principal Investigator — Meir Medical Center , Tel Aviv University
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Yes